CLINICAL TRIAL: NCT03781193
Title: Psychological Predictors of Post-surgical Recovery in Colorectal Cancer Patients: a Pilot Cohort Study
Brief Title: Psychological Predictors in Colorectal Cancer Surgery Recovery
Acronym: MIND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1945
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Cancer
Keywords: mindfulness; Psychological predictors; Colorectal surgery; ERAS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone; Perceived Stress Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires administration — Psychological and quality of life questionnaires
Other: Five Facet Mindfulness Questionnaire (FFMQ) — FFMQ is a 39-item measure consisting of five subscales (observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience).
Other: Langer Mindfulness Scale (LMS) — The LMS Tis a 21-item questionnaire, assessing four domains associated with mindful thinking: novelty-seeking, engagement, novelty producing, and flexibility.
Other: Cognitive Flexibility Scale (CFS) — The CFS is 12-item self-report test assessing awareness.
Other: Life Orientation Test (LOT) — The LOT is a 10-item, self-administered scale assessing generalized expectancies for positive versus negative outcomes.
Other: Mini Locus of Control test (MLS) — The MLS is a 6-item questionnaire that includes 3 factors : chance, powerful others, and internality.
Other: Hospital Anxiety and Depression Scale (HADS) — The HADS is a 14-items rated on a four-point Likert scale. The questionnaire was designed to screen for the presence and severity of depression (HADS-D) and anxiety (HADS-A) in people with a physical symptomatology
Other: Perceived Stress Scale (PSS) — The PSS is 14-item self-report tool commonly used to provide a global measure of perceived stress in daily life.
Other: Toronto Alexithymia Scale (TAS) — The TSA is a 20-item scale that evaluates the three components of alexithymia: difficulty to identify feelings and distinguish between feelings and bodily sensations of emotional arousal difficulty, describing feelings to others, and a cognitive style that is literal, utilitarian, and externally oriented.

SUMMARY:
This is an observation pilot trial aimed to study to the association between mindfulness and other psychological factors, including both protective and risk factors, with recovery of functional ability following colorectal cancer surgery.

DETAILED DESCRIPTION:
Preliminary evidence suggests that there are multiple variables that may influence the functional recovery following colorectal cancer surgery, some of which deal with the psychological domain. Distress and depression can negatively affect the perceptions of functional ability, while resilience and effective coping styles promote a better psychological adaptation to challenging situations. Furthermore, psychosocial prehabilitation and interventions have been proposed as a feasible and cost-effective way to positively influence the recovery after surgery in association with the Enhanced Recovery After Surgery (ERAS) protocol.

In particular, mindfulness is proved to be associated with higher quality of life in different medical conditions, including oncological patients and has been also associated with improved clinical outcomes.

The aim of the study is to investigate the association of mindfulness and other psychological predictors with functional and quality of life outcomes in patients undergoing colorectal surgery for oncological condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old (both males and females).
* Patients diagnosed with colorectal cancer.
* Patients scheduled for elective open or laparoscopic surgery for curative intent.

Exclusion Criteria:

* Patients unable to give the written informed consent.
* Patients < 18 years old.
* Patients undergoing surgery in emergency setting.
* Patients with pre-operative evidence of metastatic cancer or colorectal cancer recurrence.
* Pregnant or breastfeeding patients.
* Any condition that, in the opinion of the investigator, can interfere with the study protocol (e.g. neuropsychiatric disorders or dementia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer patients scheduled for elective curative colorectal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-03-06 (Estimated); Study Completion 2019-07-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between psychological predictors questionnaires outcome and length of hospital stay | Post-operative day 7
  Length of stay calculated in days from the day of surgery until the day of discharge
Correlation between psychological predictors questionnaires outcome and quality of life | Post-operative day 90
  Quality of Life will be assessed by using the European Organization for Research and Treatment of Cancer Quality of Life core Questionnaire (EORTC-QLQ-C30) and the European Organisation for Research and Treatment of Cancer Quality of life Questionnaire ColoRectal specific module (EORTC-QLQ-CR29)
Correlation between psychological predictors questionnaires outcome and quality of life | Post-operative month 6
  Quality of Life will be assessed by using the European Organization for Research and Treatment of Cancer quality of Life core Questionnaire (EORTC-QLQ-C30) and the European Organisation for Research and Treatment of Cancer Quality of life Questionnaire ColoRectal specific module (EORTC-QLQ-CR29)
Correlation between psychological predictors questionnaires outcome and quality of life | Post-operative month 12
  Quality of Life will be assessed by using the European Organization for Research and Treatment of Cancer Quality of Life core Questionnaire (EORTC-QLQ-C30) and the European Organisation for Research and Treatment of Cancer Quality of life Questionnaire ColoRectal specific module (EORTC-QLQ-CR29)

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- IRCCS Istituto Clinico Humanitas, Division of Colon and Rectal Surgery, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No